CLINICAL TRIAL: NCT06012006
Title: Determination of the Minimal Clinically Significant Difference (MCID) of Multidimensional Dyspnea Profile (MDP) Scores in Chronic Obstructive Pulmonary Disease (COPD) Patients During Pulmonary Rehabilitation
Brief Title: Minimal Clinically Significant Difference (MCID) of Multidimensional Dyspnea Profile (MDP) in COPD Patients Undergoing Respiratory Rehabilitation
Acronym: DYSCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP221339
Record Dates: First submitted 2023-07-24; First posted 2023-08-25 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: COPD
Keywords: Breathlessness; MCID; COPD; MDP; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulmonary rehabilitation (Experimental): COPD patients will be admitted for pulmonary rehabilitation, the duration and modalities of which vary from center to center.
  Interventions: Other: constant work-rate cycling exercise test

INTERVENTIONS:
Other: constant work-rate cycling exercise test — Description: at the end of pulmonary rehabilitation, a constant work-rate second cycling exercise test will be performed with the same duration as the cycling exercise test at inclusion

SUMMARY:
This study is designed to determine the individual threshold of minimal clinical change (MCID) for each component of the Multidimensional Dyspnea Profile (MDP) questionnaire in COPD patients undergoing pulmonary rehabilitation.

DETAILED DESCRIPTION:
The aim of the research is to determine the minimal clinically significant difference (MCID) in MDP scores in COPD patients after a respiratory rehabilitation course using the anchoring method :

* The A1 score will be compared with the Borg Affective Dyspnea (BorgA) scale.
* The sensory score will be compared with the Borg Sensory Dyspnea Scale (BorgS).
* The 5 sensory items will be compared with the Borg Sensory Dyspnea scale.
* The emotional score will be compared with the Borg Emotional Dyspnea Scale.
* The 5 emotional items will be compared with the Borg affective dyspnea scale. The various questionnaires will be administered to patients at inclusion, after a constant work-rate cycling exercise test, and at isotime during the same cycling exercise test at the end of the pulmonary rehabilitation course.

The sensitivity study will be conducted using the visual analog dyspnea scale instead of the Borg score. Finally, we will also determine the MCID using the distribution method. The MCID score will be correlated with various quality of life and physical performance scores.

ELIGIBILITY:
Inclusion Criteria:

* Gold B or D COPD patient
* Moderate to severe obstructive ventilatory disorder (FEV1<80%)
* Admitted for a pulmonary rehabilitation
* Having given free, informed and written consent

Exclusion Criteria:

* Lack of French language skills, preventing completion of questionnaires
* Cognitive impairment preventing completion of questionnaires
* Patient under guardianship
* Patient not affiliated to the social security system
* Chronic ethylism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
multidimensional (MDP) questionnaire | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  The multidimensional questionnaire measuring the sensory component of dyspnea (intensity of the 5 respiratory descriptors) and the affective component of dyspnea (immediate discomfort and intensity of emotional responses). The MDP will be carried out at the end of the constant work-rate cycling exercise test, taking into account the last 30 seconds.
sensory Borg scale | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  The two Borg scales will be carried out at the end of the constant work-rate cycling exercise test, taking into account the last 30 seconds.
affective Borg scale | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  The two Borg scales will be carried out at the end of the constant work-rate cycling exercise test, taking into account the last 30 seconds.

SECONDARY OUTCOMES:
Affective and Sensory dyspnea visual analog scale (VAS) | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  Affective and sensory dyspnea VAS will be carried out at the end of the constant work-rate cycling exercise test, taking into account the last 30 seconds.
mMRC (Modified Medical Research Council) dyspnea score | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  This 5-level score assesses the intensity of dyspnea. The consideration period will be one week.
Dyspnoea 12 | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  Multidimensional dyspnea questionnaire comprising 12 items (7 sensory and 5 affective) that can be rated from 0 (absent) to 3 (severe), i.e. a score from 0 to 36. This questionnaire measures dyspnoea over the period "these days". The consideration period will be one week
COPD Assessment Test (CAT) score | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  This questionnaire comprises 8 questions on a scale from 0 (best condition) to 5 (worst condition). The total score corresponds to the sum of the scores for each question: it ranges from 0 to 40.The consideration period will be one week.
Hospital Anxiety and Depression scale (HADS) | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  Anxiety and depression, measured by the two subscore of the HADS scale. Each subscore comprises 7 items rated from 0 (no symptoms) to 3. Seven questions relate to anxiety (total A) and seven questions relate to depression enabling us to obtain the score (maximum score = 42)The consideration period will be one week.
Saint George Respiratory Questionnaire (SGRQ) | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  evaluated by a total score and three sub-scores (symptoms, activity and impact). The total score and each sub-score are scaled from 0 to 100. The higher the score, the poorer the quality of life.The consideration period will be one week.
VQ11 | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  questionnaire consisting of 11 questions evaluated by a total score and 3 sub-scores (functional - 3 items, psychological: 4 items; relational - 4 items). Each question has 5 possible response levels, with ratings on a Likert scale ranging from 1 (not at all) to 5 (extremely). The functional, psychological and relational scores are respectively rated out of 15 for the first and 20 for the last two. The total score ranges from 11 to 55. A VQ11 total score greater than or equal to 22 reflects a patient's poor health-related quality of life.
lung function tests | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  FEV1 measurement (before and after bronchodilation), FEV1/FVC measurement, inspiratory capacity (IC) measurement, RV measurement (optional)
6 minutes walk test | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  Distance
rise chair test (optional) | at inclusion and then, up to 6 weeks (at the end of pulmonary rehabilitation course)
  number of rise

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Morelot-Panzini, MD, PhD, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal